CLINICAL TRIAL: NCT05183126
Title: Phase IV Single-arm Pharmacokinetic Study of Skeletal Muscle Area-based Paclitaxel Infusion in Patients With Cancer
Brief Title: Pharmacokinetic Study of Skeletal Muscle Area-based Paclitaxel Infusion in Patients With Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2021.109; HUM00207945 (Other: University of Michigan)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Metastatic Gastric Cancer; Esophageal Cancer
Keywords: pharmacokinetics
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Normal SMA (>7310 mm^2) (Active Comparator): Standard paclitaxel infusion time.
  Interventions: Drug: Paclitaxel
- Low SMA (5120 - 7310 mm^2) and Sarcopenic SMA (<5120 mm^2) (Experimental): Adjusted paclitaxel infusion time during only one dose; standard paclitaxel infusion time for all other doses.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Weekly intravenous (IV) infusion of a standard dose of paclitaxel 80 mg/m^2. Dose 1 is a 90-minute infusion. All other doses administered as a 1-hour infusion for a total of 12 weekly doses.
  Other Names: Taxol
  Arms: Normal SMA (>7310 mm^2)
Drug: Paclitaxel — Weekly intravenous (IV) infusion of a standard dose of paclitaxel 80 mg/m^2. Dose 1 is a 90-minute infusion.
  During doses 2-12, patients with low SMA will receive one 2-hour infusion and patients with sarcopenic SMA will receive one 3-hour infusion. All other doses during weeks 2-12 are standard infusion time.
  Other Names: Taxol
  Arms: Low SMA (5120 - 7310 mm^2) and Sarcopenic SMA (<5120 mm^2)

SUMMARY:
The primary objective of this pharmacokinetics study is to compare the maximum concentration level of paclitaxel in patients with low/sarcopenic skeletal muscle area (SMA), at the end of a 2-3 hour paclitaxel infusion, to the maximum level in patients with normal SMA at the end of a standard 1-hour infusion with the goal of determining whether lengthening the infusion in patients with low/sarcopenic SMA normalizes the levels to those of patients with normal SMA.

DETAILED DESCRIPTION:
Paclitaxel is an FDA-approved and commonly used standard of care agent for patients with early-stage breast cancer. This study will use the standard dose of 80 mg/m^2, including the typical pre-medications as per University of Michigan Rogel Cancer Center institutional standard. The only investigational component of this study is lengthening the infusion duration from 1-hour to 2 or 3 hours for a single dose in patients with low SMA.

JAN2025 update, Paclitaxel is an FDA-approved and commonly used standard of care agent for patients with early-stage breast cancer or metastatic gastric or esophageal cancers.

ELIGIBILITY:
Inclusion Criteria:

* Planned paclitaxel 80 mg/m^2, 1-hour infusion
* Evaluable computed tomography (CT) scan, positron emission tomography computed tomography (PET-CT) scan, or MRI scan (e.g. scan of the chest, abdomen, or pelvis for any indication w/in 1 year)
* Female
* ≥ 18 years old
* Adequate organ function to receive paclitaxel treatment as defined in the protocol
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Concomitant administration of any moderate or strong inducer or inhibitor of CYP2C8, including rifampin or clopidogrel.
* History of hypersensitivity reaction to paclitaxel or any components of paclitaxel (e.g., Cremophor EL) that precludes continued treatment with standard dose and infusion length
* Pregnant or nursing
* Receiving any other dose (i.e., not 80 mg/m2) or infusion rate (i.e., not 60 minute infusion) either due to toxicity during a previous cycle or any other reason

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of paclitaxel plasma | Up to week 12
  Compare Cmax in patients with lower SMA with an adjusted infusion duration (i.e., 2-hour or 3-hour) to that of patients with normal SMA receiving standard 1-hour infusion. Blood samples for pharmacokinetic analysis will be collected within 5 minutes prior to the end of SMA-based and standard paclitaxel infusions. Measurement of plasma paclitaxel concentration for Cmax will be conducted using a liquid chromatography/mass spectroscopy assay.

SECONDARY OUTCOMES:
Two- to three-hour Cmax vs. one-hour Cmax in low SMA patients | Up to week 12
  To compare Cmax in patients with lower SMA when receiving adjusted infusion duration (i.e., 2-hour or 3-hour) versus standard 1-hour infusion. Blood samples for pharmacokinetic analysis will be collected within 5 minutes prior to the end of SMA-based and standard paclitaxel infusions. Measurement of plasma paclitaxel concentration for Cmax will be conducted using a liquid chromatography/mass spectroscopy assay.
One-hour Cmax in normal SMA patients vs. one-hour Cmax in low SMA patients | Up to week 12
  To compare Cmax in patients with lower SMA versus patients with normal SMA receiving when both receive standard 1-hour infusion. Blood samples for pharmacokinetic analysis will be collected within 5 minutes prior to the end of standard 1-hour paclitaxel infusions in both groups. Measurement of plasma paclitaxel concentration for Cmax will be conducted using a liquid chromatography/mass spectroscopy assay.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L Hertz, PharmD, PhD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No